CLINICAL TRIAL: NCT02956018
Title: Continuous Monitoring of Kidney Transplant Perfusion Using Near Infra-red Spectroscopy
Brief Title: Kidney Transplant Monitoring Using Near Infra-red Spectroscopy
Status: Completed | Type: Observational
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 16HM06; 213885 (Other: IRAS)
Record Dates: First submitted 2016-11-02; First posted 2016-11-04 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Kidney Transplant; Complications
Keywords: children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Kidney transplant thrombosis (loss of blood flow) is responsible for up to 35% transplant failures in children. Detection of kidney transplant thrombosis currently relies on recognition of deterioration in parameters such as urine output and blood creatinine levels, which change relatively slowly. Confirmation is then required with an ultrasound scan. There is inherent delay in the above process, during which time some or all of the transplant kidney tissue can die, which can result in failure of the transplant.

Near infrared spectroscopy (NIRS) is a non-invasive technique used in continuous monitoring of oxygen levels in several organ systems including the brain, muscles, gut, liver and native kidneys. We hypothesise that NIRS can be applied to monitor kidney transplant blood flow in real time.

We aim to test the use of NIRS in detecting blood flow in established kidney transplants in children, and to compare it with ultrasound, the current gold standard measurement. Existing NIRS equipment would be used within its CE marked purpose measuring oxygen levels; this mechanistic study would extrapolate measured oxygen levels to determine blood flow. Participating children attending outpatient clinic for routine transplant ultrasound scans will have NIRs monitoring for a 10 minute period. NIRs data will be compared to a validated perfusion score from ultrasound images.

If this study is successful, NIRS could provide continuous monitoring of kidney transplant blood flow in the postoperative period, thus allowing immediate detection of blood flow problems. This has potential to reduce kidney transplant failures from thrombosis.

DETAILED DESCRIPTION:
The purpose of this mechanistic pilot study is to determine whether existing NIRS equipment, used within its intended CE marked purpose measuring tissue oxygenation, can reliably determine blood flow in established kidney transplants.

Objectives

1. To compare NIRS to the current gold standard measure of kidney transplant perfusion, Doppler ultrasound, in established kidney transplants in children
2. To determine the practicality of using NIRS to measure perfusion in children with established kidney transplants

Outcomes Primary Outcome • Correlation of NIRs perfusion data with Doppler ultrasound perfusion parameters assessed using a validated scale.

Secondary outcomes

• Quality of NIRS data obtained (assessed by proportion of valid readings vs lost readings)

Study Design For participating patients undergoing routine clinical outpatient renal transplant ultrasound examinations, NIRS data will be recorded on the same day. Ultrasound examinations will be undertaken by an experienced member of the radiology team following a standard protocol. NIRS data will be recorded by a member of the study team.

The ultrasound operator will perform doppler ultrasound assessment of graft parenchymal perfusion, and mark on the skin positions of the transplant upper, inter and lower poles. The ultrasound assessment will include a measurement of the distance from skin to the corticomedullary junction of the upper, inter and lower poles of the kidney transplant. NIRS data will then be recorded for 2 minutes with two NIRS sensors placed over the transplant mid and lower poles as per markings from ultrasound.

Data Collection NIRS data will be stored electronically on a password protected NHS computer and identified via an individual study number.

Oximetry readings will be exported to a password protected NHS computer for analysis. Continuous sampling data will be transformed to area under the curve (AUC) for time periods of 15 seconds, 30 seconds, 1 minute, 5 minutes and 10 minutes.

Ultrasound Doppler perfusion data will be recorded on data collection sheets labelled with the participant's study number. Data recorded will include

1. Resistive index
2. Global assessment of graft perfusion as per validated scale outlined below
3. Doppler waveform characteristics
4. Transplant parenchymal abnormalities

Renal allograft Doppler perfusion scale:

Score Doppler ultrasound assessment 0 Unidentifiable vessels

1. Few vessels in the vicinity of the hilum
2. Hilar and interlobar vessels in most of the renal parenchyma
3. Renal vessels identifiable until the arcuate arteries in the entire field of view

Data Protection Data will be collected and retained in accordance with the Data Protection Act 1998.

For identification purposes, patients' study numbers, name and hospital numbers will be stored on a single password protected NHS computer in a password protected database.

Storage of records Study documents (paper and electronic) will be retained in a secure location during and after the trial has finished. All source documents will be retained for a period of five years following the end of the study. Where trial related information is documented in the medical records - those records will be identified by a 'Do not destroy before dd/mm/yyyy' label where date is five years after the last patient last visit.

Statistical analysis

NIRS perfusion data at the time of each Doppler ultrasound will be interrogated. Continuous sampling data will be transformed to area under the curve (AUC) for time periods of 15 seconds, 30 seconds, 1 minute, 5 minutes and 10 minutes.

NIRS AUC data will be compared to Doppler ultrasound perfusion data using Spearman's correlation. Accounting for the repeated measurements within patients, mixed effects logistic regression analysis will be conducted and reciever operating characteristic curves will be determined for each NIRS AUC interval (i.e. 15 sec, 30 sec, 1,5 and 10 min), using the dichotomous Doppler ultrasound outcome as the gold standard. NIRs AUC data for perfused and non-perfused allograft poles will be compared using mixed effects regression analysis. Distributional assumptions will be investigated and where appropriate suitable transformations will be used.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 - 18 years who received kidney transplants at Great Ormond Street Children's Hospital.

Exclusion Criteria:

* patients with transplant wound complications

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 50 children with established kidney transplants undergoing follow up at Great Ormond Street Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Correlation of NIRs perfusion data with Doppler ultrasound perfusion parameters assessed using a validated scale | 6 months

SECONDARY OUTCOMES:
Quality of NIRS data obtained | 6 months
  proportion of valid readings vs lost readings

CONTACTS AND LOCATIONS:
Locations (1):
- Great Ormond Street Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No